CLINICAL TRIAL: NCT03022006
Title: Safety and Effect of Elbasvir/Grazoprevir Combination Therapy in Hemodialysis Patients With Chronic Hepatitis C
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norte Study Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Goki Suda, assistant professor, Norte Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 016-0273
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — elbasvir-grazoprevir drug combination

ARMS (1):
- Dialysis patients with genotype 1 HCV infection (Other): elbasvir/grazoprevir
  Interventions: Drug: elbasvir, grazoprevir

INTERVENTIONS:
Drug: elbasvir, grazoprevir

SUMMARY:
The number of hemodialysis patients with chronic renal failure in Japan exceeds 0.3 million and is showing an increasing trend. The rate of infection with hepatitis C virus (HCV) is high in hemodialysis patients, and it has been revealed that the prognosis is poorer in HCV-infected hemodialysis patients compared to uninfected patients; therefore, aggressive therapeutic intervention is required.Investigator previously reported the efficacy and safety of a NS5A inhibitor; daclatasvir and a HCV protease inhibitor; asunaprevir combination therapy for Japanese dialysis patients with genotype 1 HCV infection. However, the duration of the treatment is 24 week, which is quite longer than current standard 12 week therapy .

elbasvir/grazoprevir combination therapy is oral anti-HCV 12 week therapy without the use of IFN/ribavirin, and a good therapeutic effect has been reported in Japanese phase II studies . Of note is that these drugs are metabolized mainly in the liver and thus they can be used in patients with chronic renal failure. Recently, David Roth et al reported that the efficacy and safety of elbasvir/grazoprevir combination therapy for patients with hepatitis C virus genotype 1 infection and stage 4-5 chronic kidney disease. In this report, they revealed that elbasvir/grazoprevir combination therapy could achieve SVR rate of 99% in the modified full analysis set.

However, no adequate clinical investigation has been performed in Japan, thus far concerning the therapeutic effect and safety of elbasvir/grazoprevir combination therapy in Japanese hemodialysis patients.

ELIGIBILITY:
Inclusion criteria

* Patients aged 20 years or older at the time of consent
* Patients who received an adequate explanation prior to the study and provided written consent for participation in the study
* Hemodialysis patients complicated by chronic hepatitis C who have HCV Genotype 1b infection and do not meet the exclusion criteria listed in the following section

Exclusion criteria

* Patients with a past history of hypersensitivity to HCV protease inhibitors and NS5A inhibitors
* Patients with serious liver dysfunction (Child-Pugh Class B or C)
* Patients with difficult-to-control heart disease (e.g., myocardial infarction, heart failure, and arrhythmia)
* Patients who have malignant tumors, including hepatoma, at the start of treatment
* Patients on treatment with drugs listed in the contraindications for coadministration in the package insert (e.g., some antifungals, some antiepileptics, and human immunodeficiency virus (HIV) protease inhibitors)
* Patients with albumin <3.0 g/dL and platelets <75,000 /μL
* Other patients judged to be inappropriate to participate in the study by the primary physician
* Other patients judged to be inappropriate as study subjects by the study manager

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-15 (Actual); Primary Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) rate at follow-up week 12. | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Goki Suda, Dr, Principal Investigator — Norte Study Group; Naoya Sakamoto, Prof, Study Director — Norte Study Group
Locations (1):
- Hokkaido University, Sapporo, Hokkaido, Japan